CLINICAL TRIAL: NCT02200406
Title: An Open-Label Pilot Study of Desvenlafaxine for Opioid-Dependent Patients With Comorbid Depression
Brief Title: Desvenlafaxine in Opioid-Dependent Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WI187002; Pfizer Reference Award Number (Other Grant/Funding Number: WI187002)
Record Dates: First submitted 2014-07-22; First posted 2014-07-25 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2017-08

CONDITIONS: Depression; Opioid Dependence; Methadone Treatment
Keywords: Desvenlafaxine; Opioid-dependent; Addiction; Depression; Methadone; Comorbidity
MeSH Terms: conditions — Depression; Opioid-Related Disorders; Behavior, Addictive | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Desvenlafaxine (Other): * Open-label pilot study
  * Desvenlafaxine will be administered during 56 consecutive days
  * Desvenlafaxine will be administered in the morning at a 50 mg dose during weeks 1 and 2, and at 50-100 mg doses (based on the study psychiatrist's judgment) during the 6 following weeks.
  Interventions: Drug: Desvenlafaxine

INTERVENTIONS:
Drug: Desvenlafaxine — All subjects will receive 50 mg of the medication during week 1 and 2, then 50-100 mg (based on the psychiatrist judgment) for the following 6 weeks. Subjects who experience significant adverse reactions with the 100mg dose during weeks 2 to 4 could return to the lower dose of 50 mg if judged clinically appropriate by the study psychiatrist.
  Other Names: PRISTIQ

SUMMARY:
Background: Although substitution therapy has been shown to be highly effective to retain opioid-dependent patients in treatment and reduce drug use, this population is afflicted by numerous conditions including depression. Unfortunately, studies published thus far have reported inconsistent or no difference in response between placebo therapy and antidepressants such as selective serotonin reuptake inhibitors. Objective: To assess the feasibility of Desvenlafaxine (DESV) administration among opioid-dependent subjects and explore its effect on depressive symptoms. Methods: Open-label pilot trial of 8 weeks of DESV 50-100 mg/day in 20 methadone-maintained individuals with comorbid depressive symptoms at the Centre hospitalier de l'Université de Montréal. Significance: This pilot study will lay down the foundation on which a larger multisite clinical trial could be conducted to examine DESV as new treatment for opioid-dependent population with comorbid depression.

DETAILED DESCRIPTION:
To assess the feasibility, tolerability and acceptability of 8 weeks of Desvenlafaxine (DESV) administration among opioid-dependent subjects in a methadone-maintenance program, we will collect detailed information on compliance to DESV treatment, side effects, methadone plasma levels, methadone dose changes and QTc measures.

To explore the effects of DESV on depressive symptoms among opioid-dependent subjects on methadone-maintenance treatment. The severity and symptoms of depression will be evaluated by using the MADRS, the HRDS, and the CGI scale.

To explore the effects of DESV on substance use, anxiety, craving, quality of life and suicidal risk.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-TR criteria for opioid dependence;
* Subject is on methadone treatment in the substitution program for at least 4 weeks;
* Subject is aged between 18 and 65 years old;
* subject meets the DSM-V TR criteria for major depressive episode, according to the study psychiatrist and confirmed by the Mini International Neuropsychiatric Interview (MINI);
* Subject reports a score of 20 or higher on the MADRS;
* Subject is eligible for and consents to the study;
* subject is able to give valid, informed consent;
* subject is able to speak and read French or English (grade-nine level of language required)

Exclusion Criteria:

* Unstable medical illness, defined as any medical illness which has not been well-controlled with standard-of-care medications;
* Severe psychiatric condition (e.g., current acute psychosis, past or current hypomania/mania) based on the MINI;
* Pregnancy or breastfeeding;
* Inability to use a medically acceptable form of contraception throughout the study duration. A medically acceptable form of contraception is either: (1) contraceptive pill or intrauterine device or depot hormonal preparation (ring, injection, implant); and/or (2) a barrier method of contraception such as diaphragm, sponge with spermicide or condom;
* Subject currently takes another antidepressant;
* Treatment with Desvenlafaxine at any time in the past;
* Known hypersensitivity to venlafaxine;
* Subject is undergoing psychotherapies for current depression (support therapy or counseling are allowed);
* Subject failed to respond to two or more Health-Canada-approved antidepressants during current episode;
* Unstable Axis-II personality disorder or other Axis-II disorder which has been the primary focus of treatment in the past 3 months, as ascertained by a study psychiatrists;
* Medical diagnosis of kidney and/or liver failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Tolerability: Systematic Assessment for Treatment Emergent Events (SAFTEE) | 8 weeks
  Safety and adverse effects with the Systematic Assessment for Treatment Emergent Events (SAFTEE)

SECONDARY OUTCOMES:
effect of Desvenlafaxine on depressive symptoms | 8 weeks
  Responders will be determined by a 50% reduction in (Hamilton Depression Rating Scale) HAM-D scores, and remitters will be determined based on scores of ≤7.
effect of Desvenlafaxine on depressive symptoms | 8 weeks
  Responders will be determined by a 50% reduction in the Montgomery-Asberg Depression Scale (MADRS) scores, and remitters will be determined based on scores of 10.
Response to treatment | 8 weeks
  A favorable response will be defined as a score of 1 or 2 (very much or much improved) on the Clinical Global Impression CGI-I subscale
Feasibility: Proportion of persons screened who are eligible and enrolled | Baseline
  Proportion of persons screened who are eligible and enrolled
Treatment adherence | 8 weeks
  Compliance will be evaluated at each in-person follow-up visit. Treatment adherence will be calculated as the total number of tablets dispensed minus the number returned, divided by the total number of tablets dispensed
Effect of Desvenlafaxine administration on QT/QTc interval prolongation | 4 weeks
  It will be assessed by electrocardiograms (upper limit for safety should be 500ms).
Feasibility: Proportion of scheduled study visits completed and biological samples collected | 8 weeks
  Proportion of scheduled study visits completed and biological samples collected
Potential for drug interactions between methadone and antidepressants - Effect of Desvenlafaxine on methadone serum level (pharmacokinetic variability) | 4 weeks
  Change from baseline in methadone serum level. We will assessed the methadone serum level at baseline and after a month of treatment.
Methadone dose adjustments | 2 - 4 weeks
  Change from baseline in methadone dose. Each dose adjustment occurring during the trial will be noted at each follow-up visit

OTHER OUTCOMES:
Substance use | 8 weeks
  number of days of substance use as assessed with The Time Line Follow-Back (TFLB), urine-drug testing and alcohol-breathalyzer testing.
Effect of Desvenlafaxine on anxiety | 8 weeks
  Change from Baseline in anxiety and mood. It will be assessed with the Hamilton Anxiety Rating Scale (HAM-A)
Effect of Desvenlafaxine on blood pressure and heart rate | 8 weeks
  Change from Baseline in Systolic Blood Pressure and heart rate
Effect of Desvenlafaxine on opioid craving | 8 weeks
  Assessed with the abbreviated Heroin Craving Questionnaire (HCQ) - Change from Baseline in Craving.
Effect of Desvenlafaxine on quality of life | 8 weeks
  Change from baseline in Quality of life. It will be assessed with the World Health Organization Quality of Life questionnaire (WHOQOL-BREF)
Effect of Desvenlafaxine on disability | 8 weeks
  Change from baseline in disability. It will be assessed with the Sheehan Disability Scale (SDS)
Effect of Desvenlafaxine on suicidal behaviour | 8 weeks
  Change from Baseline in suicidal behaviour. It will be assessed with the Columbia-Suicide Severity Rating Scale (CSSRS)
Effect of Desvenlafaxine on testosterone level | 4 weeks
  Change from Baseline in testosterone.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Jutras-Aswad, M.D., M.Sc., Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM); Suzanne Brissette, M.D., M.Sc., Study Chair — Centre hospitalier de l'Université de Montréal (CHUM); Julie Bruneau, M.D., M.Sc., Study Chair — Centre hospitalier de l'Université de Montréal (CHUM); Paul Lespérance, M.D., M.Sc., Study Chair — Centre hospitalier de l'Université de Montréal (CHUM); Clairélaine Ouellet-Plamondon, M.D., Study Chair — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre de recherche du Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] El Hage C, Ghabrash MF, Dubreucq S, Brissette S, Lesperance F, Lesperance P, Ouellet-Plamondon C, Bruneau J, Jutras-Aswad D. A pilot, open-label, 8-week study evaluating desvenlafaxine for treatment of major depression in methadone-maintained individuals with opioid use disorder. Int Clin Psychopharmacol. 2018 Sep;33(5):268-273. doi: 10.1097/YIC.0000000000000223. PMID 29738425